CLINICAL TRIAL: NCT04639323
Title: Endoscopic Ruler for the Assessment of Variceal Bleeding Risks in Portal Hypertension (CHESS2005): A Prospective Multicenter Trial
Brief Title: Endoscopic Ruler for the Assessment of Variceal Bleeding Risks (CHESS2005)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Collaborators: LanZhou University (Other); Tianjin Second People's Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); People's Hospital of Ningxia Hui Autonomous Region (Other); The Second Affiliated Hospital of Baotou Medical College (Other); The Third Xiangya Hospital of Central South University (Other); The Second Hospital of Hebei Medical University (Other); The Affiliated Hospital Of Southwest Medical University (Other); First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, Director, Institute of Portal Hypertension, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: CHESS2005
Record Dates: First submitted 2020-11-15; First posted 2020-11-20 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Liver Cirrhosis; Portal Hypertension; Gastroesophageal Varices
Keywords: Esophagogastroduodenoscopy; Endoscopic ruler; Varices size
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overall eligible participants: Eligible participants whose varix size will be measured by endoscopists and endoscopic ruler will receive standard esophagogastroduodenoscopy
  Interventions: Diagnostic Test: Endoscopic ruler

INTERVENTIONS:
Diagnostic Test: Endoscopic ruler — Endoscopic ruler for varices in portal hypertension
  Product uses: measuring the diameter of the veins under the endoscopy for the assessment of the risk of variceal haemorrhage in patients with portal hypertension
  Black and white measuring rule is highly recognizable under the endoscopy
  The width of each cell is 1 mm, and the measuring range is 0-10 mm
  With smooth edge, safe and reliable

SUMMARY:
The presence of varices is a serious complication of portal hypertension in liver disease. To prevent variceal haemorrhage, screening and surveillance aims to detect high-risk varices related to varices size and determine the need for primary prophylaxis. Varices size evaluated by endoscopists might not be perfect reference, influenced by experience and machine. Endoscopic ruler is a novel tool to measure the varices size under the endoscopy. The investigators aim to evaluate the bias of varices size between endoscopists and endoscopic ruler as the reference.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years
* clinically evident or biopsy-confirmed cirrhosis
* Varices diagnosed by endoscopy
* written informed consent

Exclusion Criteria:

* red sign
* Active upper gastrointestinal bleeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators prospectively recruit well-defined participants with liver cirrhosis from university hospitals. Esophagogastroduodenoscopy is performed by a dedicated endoscopist at each center. Varices size is evaluated by the endoscopist and endoscopic ruler.
Sampling Method: Probability Sample
Enrollment: 266 (Estimated)
Dates: Start 2020-12-23 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
The intraclass correlation coefficient (ICC) of the varix size and the kappa value of the varices bleeding risk between endoscopists and endoscopic ruler | 2020/11/13-2022/11/13

SECONDARY OUTCOMES:
The ICC value of the varix size and the kappa value of the varices bleeding risk among endoscopists | 2020/11/13-2022/11/13
The bleeding rate of endoscopic ruler | 2020/11/13-2022/11/13
The timing of endoscopic ruler | 2020/11/13-2022/11/13
The correlation coefficient between varices size and hepatic venous pressure gradient | 2020/11/13-2022/11/13
The correlation coefficient between varices size and decompensated events | 2020/11/13-2022/11/13

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Qi, M.D., Study Chair — LanZhou University; Fengmei Wang, M.D., Principal Investigator — Tianjin Second People's Hospital; Guoxin Zhang, M.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Shengjuan Hu, M.D., Principal Investigator — People's Hospital of Ningxia Hui Autonomous Region; Xianmei Meng, M.D., Principal Investigator — The Second Affiliated Hospital of Baotou Medical College; Xiaoyan Wang, M.D., Principal Investigator — The Third Xiangya Hospital of Central South University; Zhijie Feng, M.D., Principal Investigator — The Second Hospital of Hebei Medical University; Muhan Lv, M.D., Principal Investigator — The Affiliated Hospital Of Southwest Medical University; Yiling Li, M.D., Principal Investigator — First Hospital of China Medical University
Locations (7):
- China (7):
  - The Second Affiliated Hospital of Baotou Medical College, Baotou
  - The Third Xiangya Hospital of Central South University, Changsha
  - The first hospital of Lanzhou university, Lanzhou
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin Second People's Hospital, Tianjin
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qi X, Berzigotti A, Cardenas A, Sarin SK. Emerging non-invasive approaches for diagnosis and monitoring of portal hypertension. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):708-719. doi: 10.1016/S2468-1253(18)30232-2. PMID 30215362
- [Background] Cremers I, Ribeiro S. Management of variceal and nonvariceal upper gastrointestinal bleeding in patients with cirrhosis. Therap Adv Gastroenterol. 2014 Sep;7(5):206-16. doi: 10.1177/1756283X14538688. PMID 25177367
- [Background] Bendtsen F, Skovgaard LT, Sorensen TI, Matzen P. Agreement among multiple observers on endoscopic diagnosis of esophageal varices before bleeding. Hepatology. 1990 Mar;11(3):341-7. doi: 10.1002/hep.1840110302. PMID 2312048
- [Background] Cales P, Pascal JP. Gastroesophageal endoscopic features in cirrhosis: comparison of intracenter and intercenter observer variability. Gastroenterology. 1990 Oct;99(4):1189. doi: 10.1016/0016-5085(90)90652-h. No abstract available. PMID 2203663